CLINICAL TRIAL: NCT03051139
Title: A Cluster Randomized Controlled Trial of a Multi-component Strategy to Improve Implementation of Low Tidal Volume Ventilation for Patients With Acute Respiratory Distress Syndrome
Brief Title: A Strategy to Improve Implementation of LTVV for Patients w/ ARDS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Curtis Weiss, Principal Investigator, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00202855; K23HL118139 (NIH)
Record Dates: First submitted 2016-11-28; First posted 2017-02-13 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Implementation Science; Low Tidal Volume Ventilation (LTVV)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICU A and ICU B (Experimental): This is the intervention group.
  Interventions: Behavioral: Multi-component LTVV implementation strategy
- ICU C and ICU D (No Intervention): This is the usual care group.

INTERVENTIONS:
Behavioral: Multi-component LTVV implementation strategy — Multicomponent LTVV implementation strategy consisting of: 1) physician orientation, 2) physician audit and feedback, and 3) clinical decision support comprised of a) an ARDS screening tool using a natural language processing (NLP) algorithm, b) EHR-based tasks for clinicians to complete, and c) a clinician reminder system.
  Arms: ICU A and ICU B

SUMMARY:
The primary objective of this study is to evaluate whether a multi-component implementation strategy/quality improvement intervention comprised of 1) clinical decision support that couples a natural language processing (NLP) acute respiratory distress syndrome (ARDS) recognition tool with a clinician alert system, and 2) audit and feedback improves the implementation of low tidal volume ventilation (LTVV) for patients with the acute respiratory distress syndrome (ARDS). This will be accomplished with a cluster randomized controlled trial comparing the implementation strategy to usual care

DETAILED DESCRIPTION:
Setting:

This is a multi-ICU, single-center cluster randomized trial that will be conducted among the patients and their clinicians on four adult ICU services at Northwestern Memorial Hospital. Each ICU service will act as a cluster.

Each ICU service cares for patients in one or two physical ICU locations:

* MICU service (Medical ICU location)
* NCC service (Neuroscience/spine ICU location)
* ACC service (Cardiothoracic/transplant ICU and neuroscience/spine ICU locations)
* SCC service (Cardiothoracic/transplant ICU and surgical ICU locations)

Overall Study Design:

The study will consist of a pre-trial period of baseline data collection followed by a cluster randomized controlled trial. During the pre-trial period, the investigators will retrospectively determine the proportion of patients with ARDS on each ICU service who received at least one ventilator setting adherent to LTVV in the previous one year (baseline LTVV rate). At the end of the pre-trial period, the investigators will randomize the four ICUs services into an intervention group (ICUs A and B) and usual care group (ICUs C and D). Based on pre-trial data, the investigators will calculate the difference in baseline LTVV rates between ICUs A+B and C+D, which will be used to calculate the sample size necessary for the trial period. Following the pre-trial period, ICUs A and B will begin to receive the implementation strategy while ICUs C and D will continue with usual care as a comparator group. All mechanically ventilated, non-ARDS patients on all four ICU services during the pre-trial and trial periods will also be included as a separate concurrent comparator cohort. This will allow us to assess for temporal changes in LTVV use for mechanically ventilated patients in general, and potential spill-over of LTVV use for non-ARDS patients in ICUs A and B.

Phase I: Pre-trial cohort study

The study will begin with a pre-trial cohort study. The investigators will conduct a retrospective chart review of all mechanically ventilated patients admitted to one of the four participating ICUs within the previous one year. All patients who meet the inclusion criteria as either ARDS or non-ARDS patients will be included. The main purpose of the pre-trial study is to establish a baseline rate of LTVV use in each study ICU, which will be used as part of the primary endpoint for the clinical trial described below. All secondary endpoints listed in the Appendix will be collected on all patients in the pre-trial study.

Phase II: Randomization

At the end of the pre-trial study, the investigators will randomize the four ICU services to the intervention and usual care groups. The study statistician will conduct a simple randomization approach using computer-generated random numbers to allocate each of the four ICUs to the intervention (2 ICUs) and usual care groups (2 ICUs), ensuring that there are two intervention and two usual care ICUs. The intervention ICU services will be labeled ICU A and ICU B, and the usual care ICU services will be labeled ICU C and ICU D. The allocation of each ICU will not be revealed to other study personnel until after the calculation of the baseline LTVV rates for each ICU service.

After randomization, the investigators will calculate the baseline LTVV rate in each ICU (and therefore for the intervention and usual care groups). Based on these baseline LTVV rates, the investigators will finalize the sample size calculation for the clinical trial.

Phase III: Cluster randomized controlled trial

After the randomization process is completed, the person conducting ICU randomization will reveal the allocation of ICUs to other study co-investigators. Immediately following this unblinding, the cluster randomized controlled trial will begin. The two ICUs randomized to receive usual care (ICUs C and D) will not be exposed to an intervention during the trial period. The two ICUs randomized to the intervention group (ICUs A and B) will receive the intervention for the duration of the trial period.

Implementation strategy/Intervention (ICUs A and B)

The multi-component implementation strategy/quality improvement intervention that ICUs A and B will receive during the clinical trial will consist of three parts: orientation, audit and feedback, and clinical decision support that combines an NLP-driven ARDS diagnostic screening tool, EHR-based tasks for clinicians to complete, and a clinician reminder system.

Implementation strategy component A: Orientation

The attending and fellow physicians and ICU nurse managers of ICUs A and B will be sent an email with information orienting them to the study. Respiratory therapists will not be sent the orientation email since they rotate between the different ICUs. The text of the email is shown in the Appendix (final wording may be modified).

Implementation strategy component B: Audit and feedback

Audit and feedback will be directed to ICU attendings and fellows. At the end of every ICU shift/rotation of at least five days, each physician who has cared for at least one ARDS patient in ICU A or B during the previous shift/rotation will receive an anonymous email from a study co-investigator providing their specific rate of LTVV (number of patients to whom they gave LTVV / number of ARDS patients managed).

Implementation strategy component C: Clinical decision support

The clinical decision support (CDS) intervention combines 1) an ARDS screening tool using a natural language processing (NLP) algorithm, 2) EHR-based tasks for clinicians to complete, and 3) a clinician reminder system.

1. Based on our prior research, the investigators developed a computer application that automatically screens the EHR in real-time for initial diagnostic criteria for ARDS. If a patient is flagged as meeting these initial criteria, the application will download all data necessary to make a diagnosis of ARDS according to the Berlin Definition.

   Part of the CDS intervention includes a natural language processing (NLP) program. The NLP program will analyze downloaded data and determine whether the patient has ARDS according to the Berlin Definition.
2. If a patient in ICU A or B is identified as having ARDS, the NLP program will trigger the EHR-based tasks for clinicians to complete and the clinician reminder system. The NLP will send an alert to at least one member of the study team that a patient has been identified as having ARDS.

   1. The study team member will create an order set for low tidal volume ventilation for that patient. This order set will not be signed, but will be directed to the attending and/or fellow physician to sign. The order set will include information on the patient's current tidal volume, target tidal volume for low tidal volume ventilation, and an order to initiate low tidal volume ventilation. In addition, the co-investigator will also enter a task for the patient's nurse and RT. The task will alert the nurse and RT that the patient has ARDS, and that they should discuss initiating low tidal volume ventilation with the patient's physicians.
   2. The study team member who receives the NLP alert will also send a text page to the pagers of the attending, fellow, and resident physicians currently taking care of a newly identified ARDS patient. The page will contain text suggesting that the physician consider a diagnosis of ARDS and initiate LTVV.

For all patients in ICUs A and B identified as having ARDS and reported to the co-investigator, who are subsequently not started on LTVV within 24 hours of the clinical decision support intervention described above, both the EHR-based tasks and the web pages will be repeated every 24 hours.

ELIGIBILITY:
Clinician Inclusion Criteria:

* All critical care attending physicians and critical care fellows who provide patient care on one of the participating ICU physician services at Northwestern Memorial Hospital (medical ICU [MICU], surgical critical care [SCC], anesthesia/critical care [ACC], neurocritical care [NCC]) during the study period
* All resident physicians who provide patient care on the participating ICU services during the study period
* All nurses who provide patient care in the participating ICUs during the study period
* All respiratory therapists (RTs) who provide patient care in the participating ICUs during the study period

Patient Inclusion Criteria:

* All patients admitted to a participating ICU service listed above during the study period and meeting the following additional criteria:
* Age 18 or older
* Receiving mechanical ventilation via endotracheal tube or tracheostomy
* For primary analysis: meeting Berlin Definition of ARDS (as adjudicated by NLP algorithm)(2)
* For non-ARDS comparator group: all patients meeting other inclusion criteria and not adjudicated as having ARDS
* For pre-trial period: all patients age 18 or older and receiving mechanical ventilation

Exclusion Criteria:

- Patients whose time from ARDS onset to the earlier of extubation, death, or ICU discharge is less than 24 hours. ARDS onset is defined as the time at which the latter of the following two events occurred: PaO2/FIO2 <= 300 and bilateral infiltrates reported on a chest imaging radiology report (these must be within 24 hours of each other).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06-24 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
LTVV rate | 12 months
  The primary endpoint is the difference between intervention ICUs (ICUs A and B) and usual care ICUs (ICUs C and D) in the change in the LTVV rate between the pre-trial period and the trial period. The statistical analysis of the primary endpoint will be to test the null hypothesis that there is no difference in the change in the LTVV rate between intervention and usual care groups. LTVV is defined as a patient who receives any single tidal volume less than 6.5mL/kg predicted body weight between ARDS onset and the earlier or extubation, death, or ICU discharge. ARDS onset is defined as the time at which the latter of the following two events occurred: PaO2/FIO2 <= 300 and bilateral infiltrates reported on a chest imaging radiology report, which themselves must occur within 24 hours of each other.

SECONDARY OUTCOMES:
Difference in proportions of patients receiving LTVV between intervention and usual care groups during pre-trial period | 12 months
  Difference in proportions of patients receiving LTVV between intervention and usual care groups during pre-trial period
Difference in proportions of patients receiving LTVV between intervention and usual care groups during trial period | 12 Months
  Difference in proportions of patients receiving LTVV between intervention and usual care groups during trial period
LTVV rate in individual ICUs | 12 Months
  LTVV rate in individual ICUs
Difference in overall LTVV rate between pre-trial and trial periods | 12 Months
  Difference in overall LTVV rate between pre-trial and trial periods
Percentage of time receiving LTVV | 12 Months
  Percentage of time receiving LTVV
Time from ARDS onset to LTVV initiation | 12 Months
  Time from ARDS onset to LTVV initiation
Percentage of ventilator settings adherent to LTVV | 12 Months
  Percentage of ventilator settings adherent to LTVV
ARDS duration | 12 Months
  ARDS duration
Proportion of clinicians using LTVV | 12 Months
  Proportion of clinicians using LTVV
Plateau pressure | 12 Months
  Plateau pressure
ICU and hospital length of stay | 12 Months
  ICU and hospital length of stay
ICU, hospital, 30-, 60-, 90-, 180-day and one year mortality | 12 Months
  ICU, hospital, 30-, 60-, 90-, 180-day and one year mortality
Discharge status | 12 Months
  Discharge status
Ventilator duration | 12 Months
  Ventilator duration
Intervention delivered as intended | 12 Months
  Intervention delivered as intended
Subgroup analyses of primary and secondary endpoints based on ARDS severity | 12 Months
  Subgroup analyses of primary and secondary endpoints based on ARDS severity
Subgroup analyses of primary and secondary endpoints based on FiO2 | 12 months
  Subgroup analyses of primary and secondary endpoints based on FiO2
Subgroup analyses of primary and secondary endpoints based on plateau pressure | 12 months
  Subgroup analyses of primary and secondary endpoints based on plateau pressure

CONTACTS AND LOCATIONS:
Overall Officials: Curtis H Weiss, MD, MS, Principal Investigator — Northwestern Univeristy
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No